CLINICAL TRIAL: NCT04998487
Title: A Phase 1, Randomized, Open-Label, Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous LY3471851 in Healthy Participants
Brief Title: A Single-Dose Study of LY3471851 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17604; J1P-MC-KFAL (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-08-09; First posted 2021-08-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11-15

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3471851 (Abdomen) (Experimental): LY3471851 administered subcutaneously (SC) into the abdomen.
  Interventions: Drug: LY3471851
- LY3471851 (Thigh) (Experimental): LY3471851 administered SC into the thigh.
  Interventions: Drug: LY3471851

INTERVENTIONS:
Drug: LY3471851 — Administered SC.

SUMMARY:
The main purpose of this study is to estimate how much LY3471851 gets into the blood stream and how long it takes the body to remove it when administered under the skin in healthy participants. The study will also evaluate the safety and tolerability of LY3471851. The study is expected to last up to 87 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination.
* Body weight greater than 55 kilograms (kg) and body mass index (BMI) within the range of 19 to 30 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Have evidence of clinically significant active infection, including fever 100.5ºF (38ºC) or above, within 28 days of dosing or Day 1 (before dosing)
* Have had serious, opportunistic, or chronic/recurring infection within 6 months prior to screening. Examples include but are not limited to infections requiring intravenous antibiotics, hospitalization, or prolonged treatment
* Are immunocompromised per investigator judgment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3471851 | Predose up to 56 days postdose
  PK: Cmax of LY3471851
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3471851 | Predose up to 56 days postdose
  PK: AUC of LY3471851

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (1):
- LabCorp CRU, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No